CLINICAL TRIAL: NCT02239874
Title: THE EFFECTS OF VITAMIN D ON MAMMOGRAPHIC DENSITY AND BREAST TISSUE
Brief Title: VITamin D and OmegA-3 TriaL: Effects on Mammographic Density and Breast Tissue
Acronym: VITAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rulla Tamimi, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 2014P000895; R01CA178263 (NIH)
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Benign Breast Disease
Keywords: mammographic breast density, breast disease, breast tissue
MeSH Terms: conditions — Cystic Fibrosis; Breast Diseases | interventions — Vitamin D; Fish Oils; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vitamin D placebo and fish oil placebo (Placebo Comparator): vitamin D placebo + fish oil placebo
  Interventions: Dietary Supplement: Vitamin D placebo and fish oil placebo
- Fish oil and vitamin D placebo (Active Comparator): Vitamin D placebo and 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Dietary Supplement: Fish oil and vitamin D placebo
- Vitamin D and fish oil placebo (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day and fish oil placebo
  Interventions: Dietary Supplement: Vitamin D and fish oil placebo
- Vitamin D and fish oil (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day and 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Dietary Supplement: Vitamin D and fish oil

INTERVENTIONS:
Dietary Supplement: Vitamin D and fish oil placebo — Vitamin D3 (cholecalciferol), 2000 IU per day and fish oil placebo
  Arms: Vitamin D and fish oil placebo
Dietary Supplement: Fish oil and vitamin D placebo — 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Other Names: 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Arms: Fish oil and vitamin D placebo
Dietary Supplement: Vitamin D placebo and fish oil placebo — placebo
  Arms: Vitamin D placebo and fish oil placebo
Dietary Supplement: Vitamin D and fish oil — Vitamin D3 (cholecalciferol), 2000 IU per day and 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Arms: Vitamin D and fish oil

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine whether vitamin D effects mammographic breast density, mammographic texture features, and gene expression profiles in breast biopsy tissue.

DETAILED DESCRIPTION:
Mammographic density is one of the strongest risk factors for breast cancer. It is predictive of breast cancer risk for at least 10 years in the futue and has been suggested as a surrogate marker of breast cancer risk. Several states now mandate release of mammographic density data to women. However, except for anti-hormonal therapies (e.g., tamoxifen), no interventions have been proven to reduce breast density. Thus, testing promising, well-tolerated interventions that might affect mammographic density is of substantial interest. Several lines of evidence suggest that vitamin D may play a role in breast density and breast carcinogenesis. Vitamin D reduces proliferation and promotes differentiation and apoptosis in breast cells in culture. However, no large-scale randomized studies have examined the impact of vitamin D on mammographic density. We propose to examine the randomized effects vitamin D3 on mammographic breast density in the NIH sponsored VITamin D and OmegA-3 TriaL (VITAL), an ongoing randomized, double blind, trial testing vitamin D3 (2,000 IU/day cholecalciferol) and omega-3 fatty acids (840 mg eicosapentaenoic acid [EPA]+ docosahexaenoic acid [DHA]) in the primary prevention of cancer and cardiovascular disease in a multi-ethnic population of over 24,000 men and women. In this ancillary sub study, mammograms will be obtained on 4000 women age 55-67 years (25% African-American), from baseline (pre-randomization) and after 1 and 4 years of randomized therapy. Centrally processed quantitative mammographic density and texture variation will be measured. We will determine if randomized vitamin D treatment is associated with change in mammographic features, and whether effects are modified by baseline mammographic density, and baseline 25(OH) vitamin D levels. In addition, tissue samples from women in VITAL undergoing breast biopsy/surgery, for both nonmalignant and malignant conditions, will be collected. Quantitative morphological measures, as well as gene expression assays targeting vitamin D activation and breast carcinogenesis pathways, will be performed on collected tissues among women on randomized vitamin D3 compared with placebo. This ancillary study provides a timely opportunity to test comprehensively the effects of vitamin D3 on mammographic features and breast tissue biology in a randomized setting at minimal additional cost.

ELIGIBILITY:
Inclusion Criteria:

* part of parent VITAL trial

Exclusion Criteria:

* Men,
* women with breast cancer

Ages: 55 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3894 (Estimated)
Dates: Start 2012-07; Primary Completion 2022-03 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Mammographic breast density | change baseline to 4 years
  We will collect baseline (pre-randomization), 1-year and 4-year follow-up mammograms, as well as tissue specimens from women undergoing breast biopsy/surgery for malignant and nonmalignant disease, to further elucidate the role of vitamin D on mammographic features and breast tissue biology

SECONDARY OUTCOMES:
Breast tissue | 4 years
  Quantitative morphological measures, as well as gene expression assays targeting vitamin D activation and breast carcinogenesis pathways, will be performed on collected tissues among women on randomized vitamin D3 compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Rulla M Tamimi, ScD, Principal Investigator — Brigham and Women's Hospital; Kathy Rexrode, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States